CLINICAL TRIAL: NCT06854393
Title: Lacripep, a Novel Investigational Agent, for Corneal Wound Healing and Ocular Surface Homeostasis
Brief Title: Lacripep for Corneal Wound Healing Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: TearSolutions, Inc. (Industry); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2024-0470; HT94252411092 (Other Grant/Funding Number: HJF/USAMRAA)
Record Dates: First submitted 2025-02-18; First posted 2025-03-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Corneal Epithelial Wound Healing
Keywords: Cornea; Wound healing; PRK; Lacritin; Lacripep
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Intervention Model Description: Participants will:
  1. Undergo photorefractive keratectomy (PRK), which is an eye surgery to improve vision.
  2. Use two types of experimental eyedrops three times a day for three weeks. There will be separate containers of eyedrops for the right eye and the left eye. One eye will get the active eyedrop (Lacripep) and the other eye will get the placebo eyedrop (saline).
Masking Description: Participant will receive both active treatment and placebo at the same time. One eye will receive active treatment (Lacripep) and the other eye will receive placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants will receive Lacripep in one eye and placebo in the other eye at the same time.
  Interventions: Drug: 0.00025% Lacripep ophthalmic solution and Placebo

INTERVENTIONS:
Drug: 0.00025% Lacripep ophthalmic solution and Placebo — Participant will receive Lacripep in one eye and placebo in the other eye at the same time.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of Lacripep as a therapy for superficial corneal injury repair after Photorefractive keratectomy (PRK).

DETAILED DESCRIPTION:
The purpose of this study is to assess the effect of an eyedrop medication, Lacripep, on wound healing in the cornea (the transparent tissue covering the front of the eye) such as seen after incidental or combat related trauma, or from eye surgeries like Photorefractive keratectomy (PRK). This study will help understand if Lacripep is an effective treatment in ocular surface healing and speeding visual recovery after injury.

Participants must be an active-duty service member or a dependent eligible for care at a military treatment facility.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, of any race, 21 years old and older
2. Active-duty U.S. military service members or their dependents eligible for care at Alexander T. Augusta Military Medical Center for 6-month period postoperatively
3. Desiring refractive correction of myopia up to -4.00 diopters (D) sphere with or without astigmatism 0 to -1.50 D and up to -4.00 D manifest spherical equivalent in both eyes
4. Stable refraction for the past year as demonstrated by a change in manifest refractive spherical equivalent of ≤ 0.50 diopters (D) in both eyes
5. CDVA of at least 20/20 in both eyes
6. Elected to undergo bilateral PRK
7. Able to meet follow up requirements for up to 6-month period post-operatively

Exclusion Criteria:

1. Calculated ablation depth of greater than 75 microns or other conditions in either eye which in the judgement of the investigators will require use of prophylactic MMC
2. Signs of unstable or progressive myopia, keratoconus or keratoconus suspect in either eye
3. Abnormal corneal topographic findings in either eye e.g., keratoconus, pellucid marginal degeneration
4. Treatment targeted for monovision
5. Signs and symptoms of dry eye based on: (a) Corneal fluorescein staining total score ≥4 in the National Eye Institute (NEI)/Industry Workshop scale in either eye, (b) Anethetized Schirmer test score ≤5 mm/5 minutes in either eye, (c) Symptom score ≤40 using the Symptom Assessment in Dry Eye (SANDE) questionnaire in either eye
6. Female subjects who are pregnant, breastfeeding or intend to become pregnant during the study. Pregnancy and breastfeeding are contraindications to refractive surgery in general, including PRK, whether participating in this study or not.
7. Residual, recurrent or active ocular diseases or corneal abnormalities in either eye such as iritis, uveitis, keratoconjunctivitis sicca, herpetic keratitis, vernal conjunctivitis, lagophthalmos, corneal scarring, anterior basement membrane disease, recurrent erosions, glaucoma, previous steroid responder, occludable chamber angles, visually significant cataracts
8. Previous corneal or intraocular surgery in either eye for refractive or therapeutic purposes
9. Concurrent topical or systemic medications that may impair healing, including corticosteroids, antimetabolites, isotretinoin (Accutane®), amiodarone hydrochloride (Cordarone®) and/or sumatriptan (Imitrex®) (other medications in the same family as Imitrex will still be allowed)
10. Medical condition(s), which, in the judgment of the investigator, may impair healing, including but not limited to collagen vascular disease, autoimmune disease, immunodeficiency diseases, and ocular herpes zoster or simplex.
11. Individuals not legally competent to provide informed consent (e.g., incapacitated individuals, cognitively impaired) will not be enrolled. All subjects must provide consent to participate in the study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Lacripep | Epithelial thickness assessment will be performed at 4 and 7 days postoperatively then at 1, 3 and 6 months postoperatively.
  To determine the efficacy of Lacripep for corneal wound healing, epithelial thickness will be be measured using optical coherence tomography (OCT). OCT is a non-invasive imaging technique that uses light waves to create detailed images of tissue structures.

SECONDARY OUTCOMES:
Lacripep safety | From enrollment to the end of treatment at 6 months
  To determine the safety of Lacripep, the return of corrected distance visual acuity (CDVA) will be measured using high contrast visual acuity test. Return of CDVA will be defined as percentage of eyes with no more than 1 CDVA line lost from preoperative baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary P Skurski, DO, Principal Investigator — Alexander T. Augusta Military Medical Center
Locations (1):
- Alexander T. Augusta Military Medical Center, Fort Belvoir, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yulek F, Ozdek S, Gurelik G, Hasanreisoglu B. Effect of topical steroids on corneal epithelial healing after vitreoretinal surgery. Acta Ophthalmol Scand. 2006 Jun;84(3):319-22. doi: 10.1111/j.1600-0420.2005.00632.x. PMID 16704691
- [Background] Wong HL, Poon SHL, Bu Y, Lo ACY, Jhanji V, Chan YK, Shih KC. A Systematic Review on Cornea Epithelial-Stromal Homeostasis. Ophthalmic Res. 2021;64(2):178-191. doi: 10.1159/000509030. Epub 2020 May 29. PMID 32474566
- [Background] Wolsey D, Slade S, Wirostko BM, Brandano LA, Mann BK, Durrie DS, Thompson V. Novel Cross-Linked Ocular Bandage Gel Improves Reepithelialization After Photorefractive Keratectomy: A Randomized, Masked Prospective Study. J Ocul Pharmacol Ther. 2020 Oct;36(8):602-608. doi: 10.1089/jop.2019.0156. Epub 2020 Jul 17. PMID 32701012
- [Background] Wilson SE. Interleukin-1 and Transforming Growth Factor Beta: Commonly Opposing, but Sometimes Supporting, Master Regulators of the Corneal Wound Healing Response to Injury. Invest Ophthalmol Vis Sci. 2021 Apr 1;62(4):8. doi: 10.1167/iovs.62.4.8. PMID 33825855
- [Background] Wilson SE. Corneal wound healing. Exp Eye Res. 2020 Aug;197:108089. doi: 10.1016/j.exer.2020.108089. Epub 2020 Jun 15. PMID 32553485
- [Background] Weng TH, Chang YM, Lin FH, Weng ZX, Wang TW, Chen YH, Tai MC, Chen JT, Liang CM, Lin TY. Investigation of corneal epithelial thickness and irregularity by optical coherence tomography after transepithelial photorefractive keratectomy. Clin Exp Optom. 2024 Jan;107(1):23-31. doi: 10.1080/08164622.2023.2197107. Epub 2023 Apr 20. PMID 37078178
- [Background] Weichel ED, Colyer MH, Ludlow SE, Bower KS, Eiseman AS. Combat ocular trauma visual outcomes during operations iraqi and enduring freedom. Ophthalmology. 2008 Dec;115(12):2235-45. doi: 10.1016/j.ophtha.2008.08.033. PMID 19041478
- [Background] Wang W, Despanie J, Shi P, Edman-Woolcott MC, Lin YA, Cui H, Heur JM, Fini ME, Hamm-Alvarez SF, MacKay JA. Lacritin-mediated regeneration of the corneal epithelia by protein polymer nanoparticles. J Mater Chem B. 2014 Dec 14;2(46):8131-8141. doi: 10.1039/C4TB00979G. PMID 25530855
- [Background] Wang N, Zimmerman K, Raab RW, McKown RL, Hutnik CM, Talla V, Tyler MF 4th, Lee JK, Laurie GW. Lacritin rescues stressed epithelia via rapid forkhead box O3 (FOXO3)-associated autophagy that restores metabolism. J Biol Chem. 2013 Jun 21;288(25):18146-61. doi: 10.1074/jbc.M112.436584. Epub 2013 May 2. PMID 23640897
- [Background] Wang J, Wang N, Xie J, Walton SC, McKown RL, Raab RW, Ma P, Beck SL, Coffman GL, Hussaini IM, Laurie GW. Restricted epithelial proliferation by lacritin via PKCalpha-dependent NFAT and mTOR pathways. J Cell Biol. 2006 Aug 28;174(5):689-700. doi: 10.1083/jcb.200605140. Epub 2006 Aug 21. PMID 16923831
- [Background] Vlasov A, Sia RK, Ryan DS, Mines MJ, Stutzman RD, Rivers BA, Tseng SC, Bower KS. Sutureless cryopreserved amniotic membrane graft and wound healing after photorefractive keratectomy. J Cataract Refract Surg. 2016 Mar;42(3):435-43. doi: 10.1016/j.jcrs.2015.11.045. PMID 27063525
- [Background] Vlasov A, Ryan DS, Ludlow S, Coggin A, Weichel ED, Stutzman RD, Bower KS, Colyer MH. Corneal and Corneoscleral Injury in Combat Ocular Trauma from Operations Iraqi Freedom and Enduring Freedom. Mil Med. 2017 Mar;182(S1):114-119. doi: 10.7205/MILMED-D-16-00041. PMID 28291461
- [Background] Vijmasi T, Chen FY, Balasubbu S, Gallup M, McKown RL, Laurie GW, McNamara NA. Topical administration of lacritin is a novel therapy for aqueous-deficient dry eye disease. Invest Ophthalmol Vis Sci. 2014 Jul 17;55(8):5401-9. doi: 10.1167/iovs.14-13924. PMID 25034600
- [Background] Townley R. The state of refractive surgery in the U.S. Air Force. Presented at: Military Refractive Safety and Standards Symposium; January 7-10, 2019; San Diego, CA
- [Background] Tomas-Juan J, Murueta-Goyena Larranaga A, Hanneken L. Corneal Regeneration After Photorefractive Keratectomy: A Review. J Optom. 2015 Jul-Sep;8(3):149-69. doi: 10.1016/j.optom.2014.09.001. Epub 2014 Oct 23. PMID 25444646
- [Background] Tauber J, Laurie GW, Parsons EC, Odrich MG; Lacripep Study Group; Lacripep Study Group. Lacripep for the Treatment of Primary Sjogren-Associated Ocular Surface Disease: Results of the First-In-Human Study. Cornea. 2023 Jul 1;42(7):847-857. doi: 10.1097/ICO.0000000000003091. Epub 2022 Jul 28. PMID 35942530
- [Background] Sia RK, Ryan DS, Stutzman RD, Pasternak JF, Eaddy JB, Logan LA, Torres MF, Bower KS. Wavefront-guided versus wavefront-optimized photorefractive keratectomy: Clinical outcomes and patient satisfaction. J Cataract Refract Surg. 2015 Oct;41(10):2152-64. doi: 10.1016/j.jcrs.2015.10.054. PMID 26703291
- [Background] Sridhar MS. Anatomy of cornea and ocular surface. Indian J Ophthalmol. 2018 Feb;66(2):190-194. doi: 10.4103/ijo.IJO_646_17. PMID 29380756
- [Background] Sedaghat MR, Momeni-Moghaddam H, Gazanchian M, Reinstein DZ, Archer TJ, Randleman JB, Hosseini SR, Nouri-Hosseini G. Corneal Epithelial Thickness Mapping After Photorefractive Keratectomy for Myopia. J Refract Surg. 2019 Oct 1;35(10):632-641. doi: 10.3928/1081597X-20190826-03. PMID 31610004
- [Background] Sanghi S, Kumar R, Lumsden A, Dickinson D, Klepeis V, Trinkaus-Randall V, Frierson HF Jr, Laurie GW. cDNA and genomic cloning of lacritin, a novel secretion enhancing factor from the human lacrimal gland. J Mol Biol. 2001 Jun 29;310(1):127-39. doi: 10.1006/jmbi.2001.4748. PMID 11419941
- [Background] Samudre S, Lattanzio FA Jr, Lossen V, Hosseini A, Sheppard JD Jr, McKown RL, Laurie GW, Williams PB. Lacritin, a novel human tear glycoprotein, promotes sustained basal tearing and is well tolerated. Invest Ophthalmol Vis Sci. 2011 Aug 5;52(9):6265-70. doi: 10.1167/iovs.10-6220. PMID 21087963
- [Background] Ryan DS, Sia RK, Stutzman RD, Pasternak JF, Howard RS, Howell CL, Maurer T, Torres MF, Bower KS. Wavefront-Guided Versus Wavefront-Optimized Photorefractive Keratectomy: Visual and Military Task Performance. Mil Med. 2017 Jan;182(1):e1636-e1644. doi: 10.7205/MILMED-D-15-00576. PMID 28051986
- [Background] Reynolds ME, Gu W. A new approach to categorization of ocular injury among U.S. Armed Forces. MSMR. 2022 Feb 1;29(2):8-14. PMID 35442608
- [Background] Pflugfelder SC. Advances in the diagnosis and management of keratoconjunctivitis sicca. Curr Opin Ophthalmol. 1998 Aug;9(4):50-3. doi: 10.1097/00055735-199808000-00009. PMID 10387469
- [Background] Pastor JC, Calonge M. Epidermal growth factor and corneal wound healing. A multicenter study. Cornea. 1992 Jul;11(4):311-4. doi: 10.1097/00003226-199207000-00007. PMID 1424650
- [Background] Pantalon A, Pfister M, Aranha Dos Santos V, Sapeta S, Unterhuber A, Pircher N, Schmidinger G, Garhofer G, Schmidl D, Schmetterer L, Werkmeister RM. Ultrahigh-resolution anterior segment optical coherence tomography for analysis of corneal microarchitecture during wound healing. Acta Ophthalmol. 2019 Aug;97(5):e761-e771. doi: 10.1111/aos.14053. Epub 2019 Feb 14. PMID 30762310
- [Background] Netto MV, Mohan RR, Ambrosio R Jr, Hutcheon AE, Zieske JD, Wilson SE. Wound healing in the cornea: a review of refractive surgery complications and new prospects for therapy. Cornea. 2005 Jul;24(5):509-22. doi: 10.1097/01.ico.0000151544.23360.17. PMID 15968154
- [Background] Moshirfar M, West WB Jr, Milner DC, McCabe SE, Ronquillo YC, Hoopes PC. Delayed Epithelial Healing with Corneal Edema and Haze After Photorefractive Keratectomy Using Intraoperative Mitomycin C. Int Med Case Rep J. 2021 Dec 24;14:863-870. doi: 10.2147/IMCRJ.S342774. eCollection 2021. PMID 34992474
- [Background] Mohan RR, Hutcheon AE, Choi R, Hong J, Lee J, Mohan RR, Ambrosio R Jr, Zieske JD, Wilson SE. Apoptosis, necrosis, proliferation, and myofibroblast generation in the stroma following LASIK and PRK. Exp Eye Res. 2003 Jan;76(1):71-87. doi: 10.1016/s0014-4835(02)00251-8. PMID 12589777
- [Background] Meduri A, Aragona P, Grenga PL, Roszkowska AM. Effect of basic fibroblast growth factor on corneal epithelial healing after photorefractive keratectomy. J Refract Surg. 2012 Mar;28(3):220-3. doi: 10.3928/1081597X-20120103-02. Epub 2012 Jan 9. PMID 22230058
- [Background] McKown RL, Coleman Frazier EV, Zadrozny KK, Deleault AM, Raab RW, Ryan DS, Sia RK, Lee JK, Laurie GW. A cleavage-potentiated fragment of tear lacritin is bactericidal. J Biol Chem. 2014 Aug 8;289(32):22172-82. doi: 10.1074/jbc.M114.570143. Epub 2014 Jun 18. PMID 24942736
- [Background] Klenkler B, Sheardown H, Jones L. Growth factors in the tear film: role in tissue maintenance, wound healing, and ocular pathology. Ocul Surf. 2007 Jul;5(3):228-39. doi: 10.1016/s1542-0124(12)70613-4. PMID 17660896
- [Background] Kaji Y, Obata H, Usui T, Soya K, Machinami R, Tsuru T, Yamashita H. Three-dimensional organization of collagen fibrils during corneal stromal wound healing after excimer laser keratectomy. J Cataract Refract Surg. 1998 Nov;24(11):1441-6. doi: 10.1016/s0886-3350(98)80164-8. PMID 9818332
- [Background] Li J, Lam CS, Yu M, Hess RF, Chan LY, Maehara G, Woo GC, Thompson B. Quantifying sensory eye dominance in the normal visual system: a new technique and insights into variation across traditional tests. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6875-81. doi: 10.1167/iovs.10-5549. Epub 2010 Jul 7. PMID 20610837
- [Background] Legault G. The state of refractive surgery in the U.S. Army. Presented at: Military Refractive Safety and Standards Symposium; January 7-10, 2019; San Diego, CA
- [Background] Leccisotti A. Mitomycin C in photorefractive keratectomy: effect on epithelialization and predictability. Cornea. 2008 Apr;27(3):288-91. doi: 10.1097/ICO.0b013e31815c5a51. PMID 18362654
- [Background] Laurie GW, Wang N, Raab RW, McKown RL. NFAT/mTOR signaling and downstream promotion of MUC16 expression by lacrimal prosecretory mitogen lacritin. Investigative Ophthalmology & Visual Science. 2006 May 1;47(13):1606-.
- [Background] Lau JJ, Thach AB, Burden JH, Ward TP, Hshieh PB, Hollifield RD. Eye injuries in the U.S. Armed Forces. Mil Med. 2000 Sep;165(9):683-6. PMID 11011541
- [Background] Hofmeister EM, Bishop FM, Kaupp SE, Schallhorn SC. Randomized dose-response analysis of mitomycin-C to prevent haze after photorefractive keratectomy for high myopia. J Cataract Refract Surg. 2013 Sep;39(9):1358-65. doi: 10.1016/j.jcrs.2013.03.029. Epub 2013 Jul 3. PMID 23830559
- [Background] Hofmeister E. The state of refractive surgery in the U.S. Navy. Presented at: Military Refractive Safety and Standards Symposium; January 7-10, 2019; San Diego, CA
- [Background] Heier JS, Enzenauer RW, Wintermeyer SF, Delaney M, LaPiana FP. Ocular injuries and diseases at a combat support hospital in support of Operations Desert Shield and Desert Storm. Arch Ophthalmol. 1993 Jun;111(6):795-8. doi: 10.1001/archopht.1993.01090060083028. PMID 8512480
- [Background] Hegarty DM, Carroll JR, Nguyen D, Halls VS, Robbins DI, Price TJ, Dussor G, Aicher SA. Resveratrol increases tear production and ocular pain after corneal abrasion in male, but not female, rats using a photorefractive keratectomy model. Exp Eye Res. 2022 Dec;225:109281. doi: 10.1016/j.exer.2022.109281. Epub 2022 Oct 18. PMID 36265575
- [Background] Gipson LK, Joyce NC. Anatomy and Cell Biology of the Cornea, Superficial Limbus and Conjunctiva. In: Albert DM ed. Principles and Practice of Ophthalmology third ed. Philadelphia: Saunders; 2008:423-40
- [Background] Georgiev GA, Gh MS, Romano J, Dias Teixeira KL, Struble C, Ryan DS, Sia RK, Kitt JP, Harris JM, Hsu KL, Libby A, Odrich MG, Suarez T, McKown RL, Laurie GW. Lacritin proteoforms prevent tear film collapse and maintain epithelial homeostasis. J Biol Chem. 2021 Jan-Jun;296:100070. doi: 10.1074/jbc.RA120.015833. Epub 2020 Nov 21. PMID 33187980
- [Background] Gensheimer MW, Davies MB, Ellis LC, Chou CE, Cousineau-Krieger UC, Corsini MJ, Caldwell LC, Shackelford CS. Eye trauma: Initial care (cpg id: 03). Joint Trauma System Clinical Practice Guideline. 2021. https://jts.amedd.army.mil/assets/docs/cpgs /Eye_Trauma_Initial_Care_01_Jun_2021_ID03.pdf. Accessed November 1, 2022.
- [Background] Gallagher EJ, Bijur PE, Latimer C, Silver W. Reliability and validity of a visual analog scale for acute abdominal pain in the ED. Am J Emerg Med. 2002 Jul;20(4):287-90. doi: 10.1053/ajem.2002.33778. PMID 12098173
- [Background] Fujii A, Morimoto-Tochigi A, Walkup RD, Shearer TR, Azuma M. Lacritin-induced secretion of tear proteins from cultured monkey lacrimal acinar cells. Invest Ophthalmol Vis Sci. 2013 Apr 5;54(4):2533-40. doi: 10.1167/iovs.12-10394. PMID 23482462
- [Background] Fowler WC, Chang DH, Roberts BC, Zarovnaya EL, Proia AD. A new paradigm for corneal wound healing research: the white leghorn chicken (Gallus gallus domesticus). Curr Eye Res. 2004 Apr;28(4):241-50. doi: 10.1076/ceyr.28.4.241.27837. PMID 15259293
- [Background] Fogla R, Luthra G, Chhabra A, Gupta K, Dalal R, Khamar P. Preferred practice patterns for photorefractive keratectomy surgery. Indian J Ophthalmol. 2020 Dec;68(12):2847-2855. doi: 10.4103/ijo.IJO_2178_20. PMID 33229660
- [Background] Feng MM, Baryla J, Liu H, Laurie GW, McKown RL, Ashki N, Bhayana D, Hutnik CM. Cytoprotective effect of lacritin on human corneal epithelial cells exposed to benzalkonium chloride in vitro. Curr Eye Res. 2014 Jun;39(6):604-10. doi: 10.3109/02713683.2013.859275. Epub 2014 Jan 8. PMID 24401093
- [Background] Farjo AA, Brumm MV, Soong HK. Corneal Anatomy, Physiology and Wound Healing. In: Yanoff M, Duker JS eds, Ophthalmology fourth ed. London: Elsevier; 2014:163-7
- [Background] Fantes FE, Hanna KD, Waring GO 3rd, Pouliquen Y, Thompson KP, Savoldelli M. Wound healing after excimer laser keratomileusis (photorefractive keratectomy) in monkeys. Arch Ophthalmol. 1990 May;108(5):665-75. doi: 10.1001/archopht.1990.01070070051034. PMID 2334323
- [Background] Efraim Y, Chen FYT, Cheong KN, Gaylord EA, McNamara NA, Knox SM. A synthetic tear protein resolves dry eye through promoting corneal nerve regeneration. Cell Rep. 2022 Aug 30;40(9):111307. doi: 10.1016/j.celrep.2022.111307. PMID 36044852
- [Background] Durrie DS, Wolsey D, Thompson V, Assang C, Mann B, Wirostko B. Ability of a new crosslinked polymer ocular bandage gel to accelerate reepithelialization after photorefractive keratectomy. J Cataract Refract Surg. 2018 Mar;44(3):369-375. doi: 10.1016/j.jcrs.2018.01.018. PMID 29703289
- [Background] DeLoach LJ, Higgins MS, Caplan AB, Stiff JL. The visual analog scale in the immediate postoperative period: intrasubject variability and correlation with a numeric scale. Anesth Analg. 1998 Jan;86(1):102-6. doi: 10.1097/00000539-199801000-00020. PMID 9428860
- [Background] Cockerham GC, Lemke S, Rice TA, Wang G, Glynn-Milley C, Zumhagen L, Cockerham KP. Closed-globe injuries of the ocular surface associated with combat blast exposure. Ophthalmology. 2014 Nov;121(11):2165-72. doi: 10.1016/j.ophtha.2014.06.009. Epub 2014 Aug 11. PMID 25124272
- [Background] Blanch RJ, Kerber MT, Gensheimer WG. Deployed ophthalmic workload in support of US and NATO operations in Afghanistan. BMJ Mil Health. 2021 Dec;167(6):408-412. doi: 10.1136/bmjmilitary-2019-001379. Epub 2020 Mar 5. PMID 32139414
- [Background] Buffault J, Zeboulon P, Liang H, Chiche A, Luzu J, Robin M, Rabut G, Labetoulle M, Labbe A, Baudouin C. Assessment of corneal epithelial thickness mapping in epithelial basement membrane dystrophy. PLoS One. 2020 Nov 25;15(11):e0239124. doi: 10.1371/journal.pone.0239124. eCollection 2020. PMID 33237913
- [Background] Blake CR, Cervantes-Castaneda RA, Macias-Rodriguez Y, Anzoulatous G, Anderson R, Chayet AS. Comparison of postoperative pain in patients following photorefractive keratectomy versus advanced surface ablation. J Cataract Refract Surg. 2005 Jul;31(7):1314-9. doi: 10.1016/j.jcrs.2004.11.046. PMID 16105600
- [Background] Begley C, Caffery B, Chalmers R, Situ P, Simpson T, Nelson JD. Review and analysis of grading scales for ocular surface staining. Ocul Surf. 2019 Apr;17(2):208-220. doi: 10.1016/j.jtos.2019.01.004. Epub 2019 Jan 14. PMID 30654024
- [Background] Barrientez B, Nicholas SE, Whelchel A, Sharif R, Hjortdal J, Karamichos D. Corneal injury: Clinical and molecular aspects. Exp Eye Res. 2019 Sep;186:107709. doi: 10.1016/j.exer.2019.107709. Epub 2019 Jun 22. PMID 31238077
- [Background] Bandeira F, Yusoff NZ, Yam GH, Mehta JS. Corneal re-innervation following refractive surgery treatments. Neural Regen Res. 2019 Apr;14(4):557-565. doi: 10.4103/1673-5374.247421. PMID 30632489
- [Background] Ashby BD, Garrett Q, Willcox MDP. Corneal injuries and wound healing - review of processes and therapies. Austin J Clin Ophthalmol. 2014;1(4): 1017.
- [Background] Andreotti G, Lange JL, Brundage JF. The nature, incidence, and impact of eye injuries among US military personnel: implications for prevention. Arch Ophthalmol. 2001 Nov;119(11):1693-7. doi: 10.1001/archopht.119.11.1693. PMID 11709022
- [Background] Amparo F, Schaumberg DA, Dana R. Comparison of Two Questionnaires for Dry Eye Symptom Assessment: The Ocular Surface Disease Index and the Symptom Assessment in Dry Eye. Ophthalmology. 2015 Jul;122(7):1498-503. doi: 10.1016/j.ophtha.2015.02.037. Epub 2015 Apr 8. PMID 25863420